CLINICAL TRIAL: NCT00108134
Title: A Multi-Center, Randomized, Double-Blind, Parallel-Group, Vehicle-Controlled Study to Determine the Safety of PEP005 0.0025%, 0.01% and 0.05% Gel With Two Treatment Schedules, Day 1 & 2 or Day 1 & 8 Applications to Superficial Basal Cell Carcinoma
Brief Title: Study to Determine the Safety of Two Applications of PEP005 Topical Gel to Superficial Basal Cell Carcinoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peplin (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PEP005-003; 2005/154
Record Dates: First submitted 2005-04-14; First posted 2005-04-15 (Estimated); Last update posted 2008-12-24 (Estimated); Status verified 2008-12

CONDITIONS: Basal Cell Carcinoma
Keywords: Superficial basal cell carcinoma; basal cell carcinoma; sBCC; BCC; PEP005; Topical; Dermatology
MeSH Terms: conditions — Carcinoma, Basal Cell | interventions — 3-ingenyl angelate

INTERVENTIONS:
Drug: PEP005

SUMMARY:
The purpose of this study is to determine whether topical application of PEP005 is safe for the treatment of superficial basal cell carcinoma.

DETAILED DESCRIPTION:
Basal cell carcinomas (BCCs) are a common skin problem largely caused by long term sun exposure. Current treatments include surgery, curettage/desiccation and simple excision, which are often cosmetically disfiguring. Non-invasive alternative therapy for treatment of BCC lesions is thus being researched. Sap from the plant Euphorbia peplus has been used for many years in Australia as a "folk" remedy to treat a number of skin conditions. The active component of Euphorbia peplus has been isolated and made into a gel applied directly to the skin by Peplin Ltd. To date, only one well-controlled study with PEP005 gel in humans has been completed. Sixteen patients received a single application of PEP005 0.01% or vehicle gel to actinic keratoses on the chest, shoulders, back and/or arms. Results show good tolerance and evidence of activity. The current study is designed to evaluate the safety of two applications of PEP005 gel in patients with superficial basal cell carcinoma (sBCC) on the arms, shoulders, chest, face and/or scalp, testing three concentrations according to two treatment regimens. Approximately 60 patients are planned to be included from multiple Australian centers. Efficacy and cosmetic outcome will be assessed and a recommended treatment regimen will be determined. Assignment to treatment is random and patients and medical staff will be blinded as to the treatment. Patients will have two visits for treatment application and will return for check-up visits the day after the first application and several times thereafter for approximately 3 months.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients at least 18 years of age
* One sBCC on the arm, shoulder, chest, face, neck, abdomen, leg, back or scalp suitable for surgical excision
* Histological confirmation of sBCC based on the central dermatopathologist's evaluation of the punch biopsy
* Longest pre- and post-biopsy diameter of the sBCC lesion between 4 mm and 15 mm
* Maximum thickness of 4 mm of the sBCC lesion
* Laboratory values within the reference ranges as defined by the central laboratory or "out of range" test results that are clinically acceptable to the Investigator
* Ability to follow study instructions and likely to complete all study requirements
* Written informed consent
* Male patients with a female partner of childbearing potential must use an approved form of contraception during the study and for 4 weeks after the last visit
* Agreement from the patient to allow photographs of all selected lesions (including the face) to be taken and used as part of the study data package

Exclusion Criteria:

* Location of the outside margin of the anticipated treatment area of the sBCC selected for treatment:

  1. within 10 cm of a malignant lesion that will require treatment during the study
  2. within 5 cm of an incompletely healed wound
  3. within 2 cm of a pre-malignant lesion (e.g. actinic keratosis lesion)
  4. within 2 cm of the open eyelid margins
  5. within 1 cm of a scar or an area previously treated with surgical excision
  6. on the lips
  7. on the breast
  8. on the hand or foot
  9. in a skin crease
* sBCC lesion selected for treatment requiring Mohs micrographic surgery
* Presence of known or suspected metastatic disease
* Histological evidence of actinic keratoses or nBCC in the screening visit biopsy sample
* Histological evidence of BCC with micro-nodular features or squamous metaplasia, sclerosing BCC (i.e. desmoplastic or morphoeic), or BCC with perineural involvement in the screening visit biopsy sample
* History of recurrence of the sBCC lesion
* History or evidence of skin diseases which would interfere with evaluation of the treatment area (e.g. eczema, unstable psoriasis, xeroderma pigmentosa)
* Known sensitivity to any of the ingredients in the study medication
* A cosmetic or therapeutic procedure (e.g. use of liquid nitrogen, surgical excision, curettage, dermabrasion, medium or greater depth chemical peel, laser resurfacing) within 10 cm of the selected sBCC lesion during the 3 months prior to study entry or anticipated treatment within 10 cm of the selected lesion during the study
* Treatment with 5-fluorouracil, imiquimod, diclofenac or photodynamic therapy:

  1. of lesions located within 10 cm of the selected sBCC lesion during the 3 months prior to study entry or
  2. anywhere during the 4 weeks prior to study entry or anticipated treatment during the study
* Use of acid-containing products (e.g. salicylic acids or fruit acids, such as alpha and beta hydroxy acids and glycolic acids), topical retinoids or light chemical peels within 10 cm of the selected sBCC lesion during the 3 months prior to study entry or anticipated treatment in this same area during the study
* Treatment with immuno-modulators (e.g. cyclosporine, prednisone, methotrexate, infliximab or other biological agents), cytotoxic drugs (e.g. vinblastine, cyclophosphamide, azathioprine, chlorambucil, methotrexate), or interferon/interferon inducers during the 4 weeks prior to study entry or anticipated treatment during the study
* Treatment with psoralen plus UVA or use of UVB therapy during the 6 months prior to study entry or anticipated treatment during the study
* Use of systemic retinoids (e.g. isotretinoin, acitretin) during the 6 months prior to study entry or anticipated treatment during the study
* Anticipated excessive or prolonged exposure to ultraviolet light (e.g. sunlight, tanning beds) or use of topical salves, creams or ointments to the selected lesion during the study
* Anticipated need for hospitalization or non-dermatological surgery during the study
* Concurrent disease that suppresses the immune system (e.g. HIV) or uncontrolled systemic disease (e.g. uncontrolled hypertension, poorly controlled diabetes)
* Current evidence of chronic alcohol or drug abuse
* Current enrolment in an investigational drug or device study or participation in such a study within 30 days of entry into this study
* Diagnosis of xeroderma pigmentosa or Gorlin Syndrome (i.e. Basal Cell Nevus Syndrome)
* A condition or situation which in the Investigator's opinion may put the patient at significant risk, may confound the study results, or may interfere significantly with the patient's participation in the study
* Females of child bearing potential (a female is considered of childbearing potential unless she is postmenopausal, i.e., no menses for at least 12 consecutive months, or is without a uterus)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60
Dates: Start 2005-03; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Safety

SECONDARY OUTCOMES:
Efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Greg Siller, Principal Investigator
Locations (9):
- Australia (9):
  - Southderm Pty Ltd, Sydney, New South Wales
  - St George Dermatology & Skin Cancer Centre, Sydney, New South Wales
  - Siller Medical, Brisbane, Queensland
  - Belmont Specialist Centre, Brisbane, Queensland
  - The Skin Centre, Gold Coast, Queensland
  - Skin and Cancer Foundation, Melbourne, Victoria
  - Freemantle Dermatology, Freemantle, Western Australia
  - Private Dermaology Clinic, Fremantle, Western Australia
  - St John of God Dermatology, Subiaco, Western Australia